CLINICAL TRIAL: NCT01787123
Title: Randomized, Double-blind, Placebo-controlled Pilot Trial to Investigate Safety and Efficacy of Cerebrolysin™ in Patients With Aneurysmal Subarachnoid Hemorrhage
Brief Title: Randomized, Double-blind, Placebo-controlled Trial to Investigate Safety and Efficacy of Cerebrolysin™ in Patients With Aneurysmal Subarachnoid Hemorrhage
Acronym: CESAR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kwong Wah Hospital (Other)
Responsible Party: Principal Investigator, Peter Woo Yat Ming, Associate Consultant, Kwong Wah Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CESAR Study
Record Dates: First submitted 2013-02-05; First posted 2013-02-08 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Subarachnoid Hemorrhage; Intracranial Aneurysm; Delayed Cerebral Ischemia; Delayed Ischemic Neurological Deficit
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Aneurysm | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control: standard management (Placebo Comparator): Standard management for patient suffering from aneurysmal subarachnoid haemorrhage
  Interventions: Drug: Normal Saline
- Intervention: standard management AND Cerebrolysin (Active Comparator): Standard management for aneurysmal subarachnoid hemorrhage and a 14-day administration of intravenous Cerebrolysin
  Interventions: Drug: Intravenous Cerebrolysin

INTERVENTIONS:
Drug: Intravenous Cerebrolysin — 14-day course of intravenous Cerebrolysin started within 4 days of ictus
  Arms: Intervention: standard management AND Cerebrolysin
Drug: Normal Saline — 14-day course of intravenous normal saline started within 4 days of ictus
  Other Names: Placebo
  Arms: Control: standard management

SUMMARY:
This is a randomized, placebo-controlled, single-center clinical trial investigating the effectiveness of administrating intravenous Cerebrolysin™ (EVER NEURO Pharma, Austria), a preparation of low-molecular weight neurotrophic peptides and free amino acids, in improving the functional outcome of patients suffering from aneurysmal subarachnoid haemorrhage ( SAH).

Cerebrolysin™ is a porcine-derived intravenous formulation composed of multiple lipid-soluble active agents that can cross the blood-brain barrier. It is a registered medication in several countries indicated for stroke and Alzheimer's disease. It contains several low molecular weight neuropeptides and free amino acids that possess neuroprotective and neurotrophic properties. It has been proven to arrest or mitigate several crucial steps along the ischemic cascade in preclinical studies. Cerebrolysin™ has been extensively investigated in patients suffering from Alzheimer's disease, brain trauma and ischemic stroke with promising clinical results. It's use in SAH patients has never been investigated and it is believed that it may play a role in improving clinical outcomes.

Consecutive patients aged 18 to 70 years-old diagnosed to have spontaneous subarachnoid hemorrhage secondary to a ruptured intracranial aneurysm will be randomly allocated into one of two study arms: (1) to receive intravenous Cerebrolysin™ in additional to standard of care (intervention group) or (2) to receive usual standard of care alone (control group). Permuted-block randomization will be carried out once the eligibility criteria have been fulfilled using a computer system with an allocation list of random order. Instructions on study arm allocation will be contained in sealed envelopes labeled with sequential study numbers. Patients presenting beyond 96 hours after onset of symptoms or if recruitment and randomization cannot be performed within this time period will be excluded. The reason being that post-SAH arterial vasospasm and delayed cerebral ischemia usually occurs four days after aneurysm rupture and lasts for two weeks i.e. 14 days. Should this complication arise before Cerebrolysin™ is administered there would be significant confounding of trial outcome measures . The timing of intervention is in keeping with several landmark clinical studies that have dealt with neuroprotective agents in subarachnoid hemorrhage.

Patients in the intervention group will receive in a daily total dose of 30ml of intravenous Cerebrolysin™. The study medication will be administered in three separate 10ml doses (every eight hours) diluted in 0.9% NaCl saline to a total volume of 100 ml as an intravenous infusion over a time period of 15 minutes. An identical amount of 0.9% sodium chloride (NaCl) saline (100 ml) will be used as placebo for patients allocated to the control study group. The total duration of study medication or placebo administration will be 14 days.

Cerebrolysin™ is a clear yellow solution. Since it is susceptible to photo-degeneration the preparation after dilution with 0.9% NaCl saline requires masking with a opaque plastic wrap as well as special photo-protective infusion sets. The dilution of the Cerebrolysin™ solution will be performed by ward nursing staff . Subjects in both trial groups will receive identically wrapped preparations so that both the functional outcomes assessor and patient are blind to the study arm allocation.

In addition to general demographic data, clinical data including the admission Glasgow Coma Score, severity grading of SAH, hospital stay as well as the extended Glasgow Outcome Score and modified Rankin Score upon discharge, at three months and six months will be prospectively collected. The functional outcomes assessor will be an occupational therapist unaware of the subject's trial group allocation.

Hypothesis: compared to patients receiving standard care for the management of aneurysmal subarachnoid hemorrhage alone (control), the additional administration of intravenous Cerebrolysin™ (intervention) within the acute phase of stroke is safe and improves functional outcome at six months after stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Subarachnoid hemorrhage secondary to a ruptured intracranial aneurysm confirmed by computed tomography, magnetic resonance imaging or digital subtraction angiography.
2. Any clinical grade of subarachnoid hemorrhage provided there is a reasonable prospect of survival.
3. Initiation of trial medication within 96 hours from the time of presenting symptoms.
4. Ethnic Chinese
5. Age 18-70 years-old
6. Reasonable expectation of completion of outcome measures at follow-up
7. Written informed consent

Exclusion Criteria:

1. Unsalvageable patients: fixed and dilated pupils after resuscitation or signs of brainstem herniation that precludes definitive therapy.
2. No previous history of Cerebrolysin™ exposure.
3. No known allergy to Cerebrolysin™ or porcine tissue-derived products.
4. Pregnancy or breast feeding.
5. Evidence of pre-existing major health problems
6. Suspected or known additional disease process that threatens life expectancy, for example malignancy.
7. Known or strong suspicion of drug dependency including alcohol
8. Known epilepsy
9. Any neurological or non-neurological condition independent from SAH that might influence the functional outcome or other efficacy outcome measures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Global functional performance | At six months after stroke
  Global functional performance upon discharge, at three and six months after stroke in terms of the extended Glasgow Outcome Scale (E-GOS) and modified Rankin Scale (mRS). Binary outcomes are defined as 'good/ moderate' or 'poor' in terms of these scales.
  For the E-GOS, 'good/ moderate' outcome is defined by a score of 7-8 (i.e. good recovery) and poor outcome is defined as 0-6 (i.e. moderate recovery to death). For the mRS, 'good/ moderate' outcome is defined by a score of 0-2 (i.e. asymptomatic to slight disability) and poor outcome is defined as 3-6 (moderate disability to death).

SECONDARY OUTCOMES:
Delayed ischemic neurological deficit (DIND) or delayed cerebral ischemia | At six months after stroke
Modified Barthel Index | At six months after stroke
Health Survey Short-form-12™ (SF-12™) | At six months after stroke
Mini-mental state examination (MMSE) | At six months after stroke
Neurobehavioural cognitive state examination (NCSE) | At six months after stroke
Length of hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
Cerebrolysin™-related adverse reactions | At six months after stroke
Mortality | At six months after stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Kwong Wah Hospital, Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Woo PYM, Ho JWK, Ko NMW, Li RPT, Jian L, Chu ACH, Kwan MCL, Chan Y, Wong AKS, Wong HT, Chan KY, Kwok JCK. Randomized, placebo-controlled, double-blind, pilot trial to investigate safety and efficacy of Cerebrolysin in patients with aneurysmal subarachnoid hemorrhage. BMC Neurol. 2020 Nov 3;20(1):401. doi: 10.1186/s12883-020-01908-9. PMID 33143640